CLINICAL TRIAL: NCT04893798
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, SINGLE-DOSE, PARALLEL-GROUP STUDY TO COMPARE THE PHARMACOKINETICS AND RELATIVE BIOAVAILABILITY OF MEDROXYPROGESTERONE ACETATE IN HEALTHY FEMALE PARTICIPANTS FOLLOWING SUBCUTANEOUS INJECTION OF SAYANA PRESS IN THE UPPER ARM RELATIVE TO ANTERIOR THIGH AND ABDOMEN
Brief Title: A Study Comparing Subcutaneous Injection of Sayana Press In the Upper Arm Versus Anterior Thigh and Abdomen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A6791042; 2024-513561-39-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Medroxyprogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sayana Press, Upper Arm injection (Experimental): Sayana Press, administered subcutaneously into upper arm
  Interventions: Combination Product: Sayana Press
- Sayana Press, anterior thigh (Active Comparator): Sayana Press, administered subcutaneously into anterior thigh
  Interventions: Combination Product: Sayana Press
- Sayana Press, abdomen (Active Comparator): Sayana Press, administered subcutaneously into abdomen
  Interventions: Combination Product: Sayana Press

INTERVENTIONS:
Combination Product: Sayana Press — Sayana Press is a drug-device combination and is considered a medical product in the EU.
  Other Names: Medroxyprogesterone

SUMMARY:
The purpose of the study is to compare the pharmacokinetics and relative bioavailability of medroxyprogesterone in healthy female participants following subcutaneous injection of Sayana Press into the upper arm versus anterior thigh and abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female participants, 18 to 45 years of age, inclusive, at the time of signing the ICD who are at low risk of pregnancy
* Participants who have a regular menstrual cycle (between 21 and 42 days in length).
* No previous injection of depot MPA for 1 year prior to enrollment.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* History of abnormal cervical cytology within the last 3 years that has not been adequately treated (at least 2 subsequent normal smears). However, ASCUS is permitted in this study.
* Known or suspected malignancy of the breast or genital organs.
* Known with metabolic bone disease.
* Undiagnosed abnormal genital bleeding.
* Known or suspected pregnancy; or nursing females.
* History of febrile illness within 5 days prior to the first dose.
* Participant with active thrombophlebitis or whose medical history suggests that they may be at increased risk for osteoporosis, thromboembolic disease or cerebral vascular disease.
* Use of prescription or nonprescription drugs, vitamins, herbal preparations and dietary supplements capable of inducing hepatic metabolism (eg, barbiturates, rifampicin, carbamazepine or St John's Wort) or any medication known to be a
* cytochrome P450 inhibitor within 30 days (or 5 half-lives of the substance, whichever is longer) of enrollment in the study
* Use of hormonal contraception (including hormone releasing intrauterine device) within the last 3 months (and should have resumed regular menstruation).
* Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTc interval >450 msec, complete LBBB, signs of an acute or indeterminate-age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision
* making and reporting. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding participants.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Serum Trough Concentration (Ctrough) of Medroxyprogesterone | Day 92 post dose
Area under the curve from time zero to end of dosing interval (AUCtau) | pre-dose, up to 92 days post dose
Maximum Observed Serum Concentration (Cmax) of Medroxyprogesterone | pre-dose, up to 92 days post dose

SECONDARY OUTCOMES:
Serum Progesterone Level | pre-dose, up to 99 days post dose
Serum Estradiol Level | pre-dose, up tp 99 days post dose
Serum Luteinizing Hormone (LH) Level | pre-dose, up to 99 days post dose
Serum Follicle-Stimulating Hormone (FSH) Level | pre-dose, up to 99 days post dose
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Informed consent document to 150 days post dose or until study completion, whichever is longer.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | baseline, up to 150 days post dose or until study completion, whichever is longer
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Screening, Day 1, up to 150 days post dose or until study completion, whichever is longer

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6791042